CLINICAL TRIAL: NCT04484324
Title: Optimal Duration of Stretching Exercise in Patients With Chronic Mechanical Neck Pain: A Randomized Controlled Trial
Brief Title: Optimal Duration of Stretching Exercise in Patients With Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Associate professor-chair of Physiotherapy Department Affiliation: University of Sharjah, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USharjah2020
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Mechanical Neck Pain
Keywords: Randomized controlled trial; muscle energy technique; Stretching exercises
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: A prospective, double blinded, parallel-group, randomized clinical trial was conducted at one of our university's research departments,
Who Masked: Participant, Outcomes Assessor
Masking Description: The treating therapist, for both the control and intervention groups, was unblinded to the treatment method but the subjects and assessor who conducted the measurements were blinded. Assessor blinding was obtained through an independent research assist; not knowing the study design and not specifically involved in any aspect of the tria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 60 seconds (Experimental): 60 seconds stretching group Stretching exercises for upper Trapezius and Levator the examiner will passively place the participant's head into flexion, side-bending away and rotation towards the side to be stretched (for upper trapezius muscle) and flexion, side-bending away and rotation away from the side to be stretched (for levator scapula ). The patient introduces a light resisted effort to take the stabilized shoulder towards the ear and the ear towards the shoulder. The contraction is sustained for 10 seconds and, upon complete relaxation of effort, the therapist gently eases the head/ neck into an increased degree of side-bending and rotation, where it is stabilized, as the shoulder is stretched caudally. The examiner will depress the participant's shoulder with 100 Newton's of force measured with pressure dynamometer. Once the examiner achieved this level of force, he maintains the stretch for 60 seconds . The procedure is repeated three times.
  Interventions: Other: Stretching exercises
- 30 seconds (Experimental): The same procedures while the therapist will maintain the stretch for 30 seconds.
  Interventions: Other: Stretching exercises
- 15 seconds (Experimental): The same procedures while the therapist will maintain the stretch for 15 seconds.
  Interventions: Other: Stretching exercises
- control (Placebo Comparator): The therapist maintains the same manual contact without stretching force
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Stretching exercises — Post-facilitation stretch is a technique involves a maximal contraction of the muscle at mid-range with a rapid movement to maximal length followed by a static stretch.
  Other Names: muscle energy technique

SUMMARY:
controversy remains about the stretching parameters needed to achieve a particular goal or treatment outcome. In clinical practice, multiple stretching techniques are used; nevertheless, there is no evidence-based agreement on the most effective parameters. One of these parameters, that might be affecting the treatment outcome the most, is the stretching duration, thus far there is a little agreement on the optimal stretching duration.

This non agreement in exact stretching parameters is obvious between authors and researchers in the field of muscle energy techniques (MET) as well as those who have used and advocate various durations for the passive stretch that follows the contraction phase in MET.

DETAILED DESCRIPTION:
comparison and subsequent conclusions about appropriate stretching times are mainly based on mechanical factors such as range of motion and flexibility, while ignoring the neural adversative mechanical tension that may be created during stretching exercises. According to the literature , stretching induced neural tension may adversely affect the central nervous system and nerve root function due to the absence of the perineurium, which is the primary load carrying structure. Thus, safe or unsafe limits of nerve elongation are not well established, despite several basic scientific and clinical studies.. Consequently, in the present study, the current study aimed to answer the question: Is it theoretically possible, that increased longitudinal strain and stress on the spinal cord and nerve root from continuous stretching exercises may subtly impair the neural function? Our hypothesis is that a duration threshold exists where, once reached, adverse neural function will be apparent resulting in a reduction of either or both latency and amplitudes of evoked potentials.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients had to be between 18 and 40 years of age
* have generalized neck pain for more than 3 months.
* with symptoms provoked by neck postures, movements, or palpation

Exclusion Criteria:

* Subjects' exclusion criteria included specific neck pain due to trauma, disc protrusion, whiplash, congenital deformity of the spine, spinal stenosis, neoplasm, inflammatory or rheumatic disease. Furthermore, subjects were excluded if they had a history of spine surgery and any objective findings consistent with neurological conditions and vascular disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
The change in peak-to-peak amplitudes of dermatomal somatosensory evoked potentials | will be measured at two intervals ;pre-treatment and 24 Hours after treatment
  Dermatomal Somatosensory Evoked Potentials will be elicited by repetitive, square wave (0.5 ms) electrical pulses (at 3 Hz) from standard clinical surface gel electrodes (20 mm) overlying cervical sensory dermatomes. Dermatomal somatosensory evoked potential will be collected at a stimulus intensity well above perception threshold.Complete recording runs will be undertaken during each session with averages of 250 to 1200 cortical responses from scalp surface recording electrodes (C3'-C4' in a 10-20 electrode configuration) of the contralateral scalp to the C4 to C8 dermatomes being stimulated

SECONDARY OUTCOMES:
The change in Neck Disability Index | will be measured at two intervals ;pre-treatment and 24 Hours after treatment
  The Neck Disability Index , consisting of 10 items related to daily living activities, will be our primary patient-reported outcome measure. Each item is scored out of five (with the no disability response given a score of 0) giving a total score for the questionnaire out of 50. Higher scores represent greater disability.
The change in Cervical range of motion | will be measured at two intervals ;pre-treatment and 24 Hours after treatment
  Cervical spine global range-of-motion will be measured using the valid and reliable cervical range-of-motion (CROM) device. The participant will perform flexion, extension, right/left lateral flexion, right/left rotation in upright sitting. The patient was instructed to perform each movement when he/she attained the maximum active range of motion. Three trials were conducted for each direction of movement, and the average of the three measurements will be recorded for analysis.
The change in Neck pain intensity | will be measured at two intervals ;pre-treatment and 24 Hours after treatment
  Neck pain intensity will be measured using the numerical pain rating scale . The patients will be asked to place a mark along the line indicating their current pain intensity; 0 reflecting ''no pain'' and 10 reflecting the ''worst pain''.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Moustafa, Principal Investigator — University of Sharjah
Locations (2):
- United Arab Emirates (2):
  - Ibrahim Moustafa, Sharjah city, United Arab Emirate
  - University of Sharjah, Sharjah city

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data and related data dictionaries available
Supporting Information: Study Protocol, SAP
Time Frame: After 6 months and will become available for one year
Access Criteria: not identified yet

REFERENCES:
- [Result] Allison, T, G McCarthy, C C Wood, and S J Jones. 1991. "Potentials Evoked in Human and Monkey Cerebral Cortex by Stimulation of the Median Nerve. A Review of Scalp and Intracranial Recordings." Brain : A Journal of Neurology, December, 2465-2503. Baker, P F, M Ladds, and K A Rubinson. 1977. "Measurement of the Flow Properties of Isolated Axoplasm in a Defined Chemical Environment [Proceedings]." The Journal of Physiology 269 (1): 10P-11P. http://www.ncbi.nlm.nih.gov/pubmed/70528. Bandy, William D, and Jean M Irion. 1994. "The Effect of Time on Static Stretch on the Flexibility of the Hamstring Muscles." Physical Therapy 74 (9): 845-50. https://doi.org/10.1093/ptj/74.9.845. Bandy, William D, Jean M Irion, and Michelle Briggler. 1997. "The Effect of Time and Frequency of Static Stretching on Flexibility of the Hamstring Muscles." Physical Therapy 77 (10): 1090-96. https://doi.org/10.1093/ptj/77.10.1090. Bijur, Polly E, Clarke T Latimer, and E John Gallagher. 2003. "Validation of a Verbally Administered Numerical Rating Scale of Acute Pain for Use in the Emergency Department." Academic Emergency Medicine : Official Journal of the Society for Academic Emergency Medicine 10 (4): 390-92. http://www.ncbi.nlm.nih.gov/pubmed/12670856. Breig, Alf. 1978. Adverse Mechanical Tension in the Central Nervous System: An Analysis of Cause and Effect: Relief by Functional Neurosurgery. Almqvist & Wiksell International. Chaitow, Leon., Helge. Franke, and Leon. Chaitow. 2013. Muscle Energy Techniques. Churchill Livingstone/Elsevier. Cox, James M. 2000. "A Review of Biomechanics of the Central Nervous System. Part I: Spinal Canal Deformations Caused by Changes in Posture (Multiple Letters)." Journal of Manipulative and Physiological Therapeutics. https://doi.org/10.1016/s0161-4754(00)90252-5. Cunha, ACV, TN Burke, FJR França, AP Marques - Clinics, and undefined 2008. n.d. "Effect of Global Posture Reeducation and of Static Stretching on Pain, Range of Motion, and Quality of Life in Women with Chronic Neck Pain: A Randomized Clinical." SciELO Brasil. Accessed July 21, 2020. https://www.scielo.br/scielo.php?pid=S1807-59322008000600010&script=sci_arttext&tlng=pt. "Effectiveness of a Home Program of Ischemic Pressure Followed by Sustained Stretch for Treatment of Myofascial Trigger Points." 2016. Physical Therapy, November. https://doi.org/10.1093/ptj/80.10.997. Fejer, René, Kirsten Ohm Kyvik, and Jan Hartvigsen. 2006. "The Prevalence of Neck Pain in the World Population: A Systematic Critical Review of the Literature." European Spine Journal. Springer. https://doi.org/10.1007/s00586-004-0864-4. Fernández-de-las-Peñas, César, Luis Palomeque-del-Cerro, Cleofás Rodríguez-Blanco, Antonia Gómez-Conesa, and Juan C. Miangolarra-Page. 2007. "Changes in Neck Pain and Active Range of Motion After a Single Thoracic Spine Manipulation in Subjects Presenting with Mechanical Neck Pain: A Case Series." Journal of Manipulative and Physiological Therapeutics 30 (4): 312-20. https://doi.org/10.1016/j.jmpt.2007.03.007. Grosso MJ, Hwang R, Mroz T, Benzel E, Steinmetz M P. 2013. "Relationship between Degree of Focal Kyphosis Correction and Neurological Outcomes for Patients Undergoing Cervical Deformity Correction Surgery." J Neurosurg Spine. 18 (6): 537-44. Harrison, D D E, R Cailliet, D D E Harrison, S J Troyanovich, and S O Harrison. 1999. "A Review of Biomechanics of the Central Nervous System--Part II: Spinal Cord Strains from Postural Loads." Journal of Manipulative and Physiological Therapeutics 22 (5): 322-32. http://www.ncbi.nlm.nih.gov/pubmed/10395435. Harrison, D E, R Cailliet, D D Harrison, S J Troyanovich, and S O Harrison. n.d. "A Review of Biomechanics of the Central Nervous System--Part III: Spinal Cord Stresses from Postural Loads and Their Neurologic Effects." Journal of Manipulative and Physiological Therapeutics 22 (6): 399-410. http://www.ncbi.nlm.nih.gov/pubmed/10478773. Jeffery Brent Feland Joseph William Myrer, +2 authors G W Measom. 2001. "The Effect of Duration of Stretching of the Hamstring Muscle Group for Increasing Range of Motion in People Aged 65 Years or Older." Physical Therapy, May. https://doi.org/10.1093/ptj/81.5.1110.